CLINICAL TRIAL: NCT04231071
Title: Randomized Double-blind Controlled Multicenter Trial Comparing Suture and Mesh Repair in Small Umbilical Hernias in Adults
Brief Title: Mesh Versus Suture Repair in Umbilical Hernias - A Multicenter Trial
Acronym: SUMMER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Maria Melkemichel, Medical Doctor, Resident in General Surgery, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SUMMER2020; SUMMER Trial (Other: Karolinska Institute)
Record Dates: First submitted 2020-01-10; First posted 2020-01-18 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-10

CONDITIONS: Umbilical Hernia
Keywords: Small umbilical hernias; mesh repair; suture repair; recurrence
MeSH Terms: conditions — Hernia, Umbilical; Recurrence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sutured group (Active Comparator): Controlled group: Primary suture repair of the small umbilical hernia defect
  Interventions: Device: Onlay Mesh group
- Onlay Mesh group (Experimental): Intervention group: Primary suture repair of the small umbilical hernia defects + a small Onlay mesh on the closed defect.
  Interventions: Device: Onlay Mesh group

INTERVENTIONS:
Device: Onlay Mesh group — Primary suture repair with a small only mesh on the closed defect

SUMMARY:
Umbilical hernia repair is one of the most common surgical performance in general surgery. Up to now, the use of suture repair has been the preferred technique for small umbilical hernia defects without any gold standard procedure. Mesh have been reserved to larger umbilical hernia defects. However, there is an increasing evidence that mesh reinforcement could be advantageous to lower the high recurrence rates also in smaller umbilical hernias. A remained important question is in what anatomical position the mesh should be placed. The investigators hypothesize that the use of an onlay mesh in small umbilical hernia defects can reduces recurrence rates without increasing postoperative complications compared to a suture repair.

DETAILED DESCRIPTION:
The trial is a prospective multicenter randomized clinical trial comparing onlay mesh to suture repair. Two hundred and eighty-eight patients with a primary elective umbilical hernia below and equal to 2 cm from seven Swedish participating surgical centers will be enrolled. Randomization will be performed intraoperatively following the measurement of the defect (with stratification for centra and for the defect size) to either closing the small umbilical defect with a simple primary suture repair or closing the defect with a simple primary suture repair with an attached small flat lightweight polypropylene only mesh on the aponeurosis. Trial participants, investigators and follow-up clinical surgeons will be blinded for the assigned allocation. The primary endpoint will be recurrence at 1 and 3 years. Secondary endpoint will be surgical site postoperative complications at 30 days and pain 1 year after surgery. As follows, participants will be visiting the outpatient clinical at 30 d, 1 year and 3 year after surgery.

All analyses will be performed according to the intention to treat principle and as specified in the analyses plan of the study protocol.

There is no randomized clinical trial today comparing recurrence rates between an onlay mesh repair and a suture repair for small umbilical hernia defects. The trial design allows a good detection of differences in recurrence with the large sample size and the adequate follow-up. Surgeons are becoming more aware of the mesh's advantage even for the small defects, but are reluctant to use a mesh due to anatomical positions with a large dissection and an increased risk of complications. A small onlay mesh could be an easy and safe method of choice for small umbilical hernia defects to avoid increased recurrence rates. Guidelines for small umbilical hernia repairs have stressed out the need for reliable data for treatment recommendations. The investigators can expect that the trial will have a direct implication on small umbilical hernia repair standards.

The clinical study protocol has underwent full external peer review as part of the funding process with Research funding from SLL (Stockholms läns landsting) Karolinska Institutet. Approval of the protocol by the Swedish Ethical Review Authority was obtained at December 2018 and January 2020.

ELIGIBILITY:
Inclusion Criteria

• Elective surgery of a primary umbilical hernia with a defect ≤ 2 cm that is measured clinically or with radiology.

Exclusion Criteria:

* Incisional hernia: previous surgery in the area of the operation
* Recurrent umbilical hernia
* Epigastric hernia (a defect from 3 cm below the xiphoid till 3 cm above the umbilicus) [20]
* Another operative procedure at the same time (i.e. cholecystectomy)
* An umbilical hernia with a defect > 2 cm measured clinically, with radiology or intra-operatively
* Multiple defects
* Pregnancy
* Infected wounds
* Acute operation (incarcerated hernia)
* BMI>35
* Ascites
* Immunosuppression
* Anticoagulant treatment (Warfarin, NOAK)
* Connective tissue disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Hernia recurrence rate | 3 year
  To evaluate whether an onlay mesh in the repair of primary small umbilical hernias ≤ 2 cm reduces recurrence rate compared to suture repair 3 year after surgery
Hernia recurrence rate | 1 year
  To evaluate whether an onlay mesh in the repair of primary small umbilical hernias ≤ 2 cm reduces recurrence rate compared to suture repair 1 year after surgery.

SECONDARY OUTCOMES:
Difference in Surgical postoperative complication rate | 30 days
  To compare the two groups of patients with regard to surgical postoperative complications (seroma, hematoma, infection) 30 days after surgery.
Difference in Pain rate after surgery assessed by VHPQ | 1 year
  To compare the two groups of patients with regard to postoperative pain rate 1 year after surgery assessed by VHPQ (Ventral Hernia Pain Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Björn Widhe, MD, PhD, Principal Investigator — Department of Clinical Sciences, Danderyds Hospital, Karolinska Institutet; Sven Bringman, MD, PhD, Principal Investigator — Department of Clinical Sciences, Danderyds Hospital, Karolinska Institutet
Locations (7):
- Sweden (7):
  - Enköping Lasarett, Enköping
  - Frölunda Hospital, Gothenburg
  - Mora Lasarett, Mora
  - Department of Surgery at Södertälje Hospital, Södertälje
  - Danderyds Hospital, Stockholm
  - Norrtälje Hospital, Stockholm
  - Sophiahemmet/GHP, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bergstrom M, Widhe B, Granasen G, Lof Granstrom A, Ohlsson J, Schult S, Dahlstrand U, Osterberg J, Loogna P, Bringman S, Melkemichel M. Onlay mesh versus suture repair for smaller umbilical hernias in adults-early results from SUMMER trial: randomized clinical trial. BJS Open. 2024 Dec 30;9(1):zrae173. doi: 10.1093/bjsopen/zrae173. PMID 40037347
- [Derived] Melkemichel M, Bringman S, Granasen G, Widhe B. SUMMER Trial: mesh versus suture repair in small umbilical hernias in adults-a study protocol for a prospective randomized double-blind multicenter clinical trial. Trials. 2021 Jun 22;22(1):411. doi: 10.1186/s13063-021-05366-7. PMID 34158088

DOCUMENTS (2):
  • Study Protocol (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT04231071/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT04231071/SAP_001.pdf